CLINICAL TRIAL: NCT01929512
Title: An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics After the Administration of HCP1201 Tablet 750/20 mg and Coadministration of Metformin SR 750 mg and Rosuvastatin 20 mg in Healthy Volunteers
Brief Title: Comparison of PK After Administration of HCP1201 and Co-administration of Metformin SR 750mg and Rosuvastatin 20mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MERO-103
Record Dates: First submitted 2013-08-07; First posted 2013-08-28 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HCP1201, Part 1 (Experimental): Participants received a single oral dose of the HCP1201 750/20mg under fasting condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: HCP1201 750/20mg
- Metformin and Rosuvastatin, Part1 (Active Comparator): Participants received a single oral dose of coadministration of Metformin SR 750mg and Rosuvastatin 20mg under fasting condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: Metformin SR 750mg; Drug: Rosuvastatin 20mg
- HCP1201, Part 2 (Experimental): Participants received a single oral dose of the HCP1201 750/20mg under fed condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: HCP1201 750/20mg
- Metformin and Rosuvastatin, Part 2 (Active Comparator): Participants received a single oral dose of coadministration of Metformin SR 750mg and Rosuvastatin 20mg under fed condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: Metformin SR 750mg; Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: HCP1201 750/20mg — 750mg Metformin/20mg rosuvastatin fixed dose combination tablet orally in the morning on day1 or day8.
  Arms: HCP1201, Part 1; HCP1201, Part 2
Drug: Metformin SR 750mg — Co-administration of Metformin 750mg and Rosuvastatin 20mg orally in the morning on day1 or day8.
  Other Names: Glucophage SR 750 mg
  Arms: Metformin and Rosuvastatin, Part 2; Metformin and Rosuvastatin, Part1
Drug: Rosuvastatin 20mg — Co-administration of Metformin 750mg and Rosuvastatin 20mg orally in the morning on day1 or day8.
  Other Names: Crestor 20mg
  Arms: Metformin and Rosuvastatin, Part 2; Metformin and Rosuvastatin, Part1

SUMMARY:
To compare the pharmacokinetic characteristics between HCP1201 tablet 750/20 mg and co-administration of metformin 750 mg plus rosuvastatin 20 mg under fasted and fed state, respectively.

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics After the Administration of HCP1201 Tablet 750/20 mg and Coadministration of Metformin SR 750 mg and Rosuvastatin 20 mg in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age 20~55 years
2. The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
3. Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
4. Subject who has the ability and willingness to participate the whole period of trial

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Glomerular filtration rate is under 60ml/min which is calculated by serum creatinine value.
3. Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.
4. SBP: lower than 90mmHg or higher than 150mmHg, DBP: lower than 60mmHg or higher than 100mmHg
5. History of relevant drug allergies or clinically significant hypersensitivity reaction.
6. History of drug abuse or positive drug screening.
7. Participation in other drug studies within 60days prior to the drug administration.
8. Whole blood donation within 60 days, blood component donation within 30 days or who got transfusion within 30days.
9. Subjects who took prescription drugs within 14 days from the patient screening or non-prescription medicine within 7 days which can affect the result of this clinical trial (acceptable according to the investigator's judgement)
10. Subjects who took medicines(e.g. proton pump inhibitor, rifampicin, oriental medicines, etc.) within 30days that can affect absorption, distribution, metabolism, elimination of metformin/rosuvastatin.
11. Intake of more than 140g of alcohol per week or who can't abstain from alcohol during the trial.
12. Subjects who smoke more than 10 cigarettes per day or who can't quit smoking during the trial.
13. Positive screening on Hepatitis B surface antigen(HBsAg), anti-Hepatitis C virus(HCV) or anti-Human immunodeficiency virus(HIV).
14. Genetic myopathic disorder or related family history, medical history of myopathic disorder caused by medication.
15. Clinically inappropriate laboratory test result.
16. Clinically inappropriate electrocardiogram result.
17. Subjects who judged ineligible by the investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
metformin, rosuvastatin Cmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
metformin, rosuvastatin AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

SECONDARY OUTCOMES:
Metformin, rosuvastatin Tmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin T1/2 | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin AUCinf | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin CL/F | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin Vd/F | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

CONTACTS AND LOCATIONS:
Overall Officials: JaeWook Ko, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea